CLINICAL TRIAL: NCT03433300
Title: Do Microprocessor Knees Improve Outcomes in Early Prosthetic Rehabilitation Compared to Nonmicroprocessor Knees?
Brief Title: Microprocessor Knees in Early Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); Otto Bock Healthcare Products GmbH (Industry)
Responsible Party: Principal Investigator, Sara Morgan, Acting Assistant Professor, Department of Rehabilitation Medicine, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00003524
Record Dates: First submitted 2018-02-08; First posted 2018-02-14 (Actual); Last update posted 2020-09-11 (Actual); Status verified 2020-09

CONDITIONS: Amputation

STUDY DESIGN:
Intervention Model Description: Pilot randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: Investigators who will conduct performance-based assessments will be blinded to the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Microprocessor Knee (Experimental): Ottobock Kenevo/Ottobock C-Leg
  Interventions: Device: Ottobock Kenevo/C-Leg
- Nonmicroprocessor knee (Active Comparator): Ottobock 3R60 for K3 participants, Ottobock 3R62 for K2 participants.
  Interventions: Device: Ottobock 3R60/3R62

INTERVENTIONS:
Device: Ottobock Kenevo/C-Leg — Microprocessor-controlled prosthetic knee
  Arms: Microprocessor Knee
Device: Ottobock 3R60/3R62 — Nonmicroprocessor-controlled knee
  Arms: Nonmicroprocessor knee

SUMMARY:
High-quality, empirical evidence to guide prosthetic rehabilitation following amputation ensures that Service members, Veterans, and civilians who experience limb loss have the potential to receive the highest quality care, regain mobility, return to gainful employment, and reintegrate into their communities. However, evidence to inform prosthetic care during the crucial post-amputation period is extremely limited. The proposed research will address this gap in knowledge by evaluating functional and patient-centered health outcomes associated with use of two distinct prosthetic knee technologies in early rehabilitation following transfemoral amputation. This novel, comparative effectiveness research aligns with the Prosthetic Outcomes Research Award (PORA) focus area of understanding the management of patient rehabilitation strategies throughout the rehabilitation process following neuromuscular injury.

The long-term goals of this project are to optimize early rehabilitation processes and associated outcomes for Service members, Veterans, and civilians with lower limb amputation. The purpose of this study is to evaluate the potential for different prosthetic knee technologies to promote function, health, and quality of life following amputation. A pilot randomized controlled trial will be conducted to compare falls, step activity, balance confidence, mobility, health-related quality of life, and community integration of people with recent transfemoral amputation in two prosthetic knee conditions: a microprocessor knee (MPK) with control of stance phase and a non-microprocessor knee (NMPK) that is appropriate for people in early rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older, Unilateral transfemoral amputation, Between 4-16 weeks post amputation, Deemed ready for prosthetic fitting by a physician, No current or prior transfemoral prosthetic use, Able to read, write and communicate in English, Weight 125kg (275lbs) or less

Exclusion Criteria:

* Diagnosis of health condition (i.e. advanced cardiac disease, severe or end-stage pulmonary disease or severe dementia) that prevents safe prosthesis use or community ambulation with prosthesis, Weight greater than 125kg (275lbs)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2018-04-13 (Actual); Primary Completion 2020-05-15 (Actual); Study Completion 2020-05-15 (Actual)

PRIMARY OUTCOMES:
Prosthetic Limb Users Survey of Mobility | Monthly for 3 months
  Self-reported prosthetic mobility

SECONDARY OUTCOMES:
Fall frequency | Monthly for 3 months
  Number of falls while using the prosthesis
Daily step count | Average daily step count by month for 3 months
  Walking activity measured with StepWatch Monitor
Timed up and go | Monthly for 3 months
  Timed performance test that measures rising from a chair, walking 3m, and returning to a seated position.
Amputee Mobility Predictor (AMPPro) Assessment Tool | Monthly for 3 months
  The name of this tool is the Amputee Mobility Predictor (AMPPro) and it was developed by Robert Gailey, PhD, PT (https://www.sralab.org/rehabilitation-measures/amputee-mobility-predictor-0). The AMPPro assesses performance-based mobility for people who use prosthetic limbs. Example items include standing balance, ability to vary cadence, and ability to step over an obstacle.
Six-minute walk test | Monthly for 3 months
  Evaluates distance walked over 6 minute time frame with rest as needed
Gait quality | Monthly for 3 months
  GaitRite System, pressure sensitive instrumented walkway will collect average walking speed, step width, step time asymmetry during 6 minute walk test
Activities-Specific Balance Confidence Scale (ABC) | Baseline and monthly for 3 months
  The Activities-Specific Balance Confidence Scale (ABC) measures the construct of balance confidence. The 16-item ABC survey asks respondents to rate their confidence in performing a variety of activities without becoming unstable (e.g., walking in the home, walking on a ramp, walking in crowds). Response options range from "no confidence" to "completely confident" when performing the activity. The revised scale proposed by Sakakibara (2011) will be used to calculate a total balance confidence score; scores for participants will range from 0 (low balance confidence) to 4 (high balance confidence).
Patient Reported Outcomes Measurement Information System 29-item profile (PROMIS-29) version 1.0 | Baseline and monthly for 3 months
  Self-reported measure of Physical Function, satisfaction with social roles, fatigue, sleep disturbance, pain intensity, pain interference, anxiety and depression
Reintegration to Normal Living Index (RNLI) | Baseline and monthly for 3 months
  11 item questionnaire to assess self-reported physical, social and psychologic performance following injury

CONTACTS AND LOCATIONS:
Overall Officials: Sara J Morgan, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No